CLINICAL TRIAL: NCT04603677
Title: Northern Colorado Coronavirus Biobank: A Biorepository for Acute and Convalescent Patient Samples From Coloradoans Infected With SARS-CoV-2 (Severe Acute Respiratory Syndrome-Coronavirus-2)
Brief Title: Northern Colorado COVID-19 Biobank
Acronym: NoCo-CoBio
Status: Completed | Type: Observational
Sponsor: Colorado State University (Other)
Collaborators: University of Colorado Health (Other)
Responsible Party: Principal Investigator, Elizabeth P Ryan, Associate Professor, Colorado State University
Other Study IDs: 20-10063H
Record Dates: First submitted 2020-10-25; First posted 2020-10-27 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Covid19
Keywords: biobank; biorepository; SARS-CoV-2 infection; COVID-19; coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, stool, saliva, nasopharyngeal swab specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute phase of SARS-CoV-2 infection: Participants with an acute SARS-CoV-2 infection. Intervention will not be implemented in this study.
- Convalescent phase of SARS-CoV-2 infection: Participants with a previous diagnosis of SARS-CoV-2 infection, now in the convalescent phase of disease. Intervention will not be implemented in this study.

SUMMARY:
The NoCo-CoBio Project is a biobanking effort to store and preserve saliva, nasopharyngeal, stool and blood specimens from SARS-CoV-2 PCR (polymerase chain reaction) positive individuals.

DETAILED DESCRIPTION:
The investigators have created a biorepository of stool, saliva, nasopharyngeal swab specimens, peripheral blood mononuclear cells, serum, and plasma from SARS-CoV-2 infected individuals for research purposes. The multifaceted biorepository will be used to establish markers predicting various presentations of COVID-19 (coronavirus disease 2019).

ELIGIBILITY:
Inclusion Criteria:

* Those who have had a positive SARS-CoV-2 PCR test

Exclusion Criteria:

* under 18 years of age
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators aim to enroll individuals who have had a positive SARS-CoV-2 PCR, with a goal of enrolling 100 hospitalized patients with acute SARS-CoV-2 infection, as well as 100 convalescent participants.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of parameters for markers of SARS-CoV-2 infection and predictors for severe disease | 6 months
  Evaluation of parameters for markers of SARS-CoV-2 infection and predictors for severe disease

SECONDARY OUTCOMES:
Evaluation of markers and predictors of post acute sequelae of COVID-19 | 2 years
  Evaluation of markers and predictors of post acute sequelae of COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Baxter, Study Director — Colorado State University
Locations (4):
- United States (4):
  - Colorado State University, Fort Collins, Colorado
  - Poudre Valley Hospital, UCHealth, Fort Collins, Colorado
  - Greeley Hospital, UCHealth, Greeley, Colorado
  - Medical Center of the Rockies, UCHealth, Loveland, Colorado

REFERENCES:
- [Derived] Whitcomb LA, Berry K, LaVergne SM, Natter N, Baxter BA, Rao S, Tipton M, Gritsenko MA, Weitz KK, Gerbasi V, Bramer LM, Piehowski PD, Webb TL, Henao-Tamayo M, Chicco AJ, Dunn J, Dutt TS, Ryan EP. Blood pro-thrombotic analytes and platelet activation are associated with post-acute sequelae of COVID-19. BMC Infect Dis. 2025 Dec 10;26(1):61. doi: 10.1186/s12879-025-11824-3. PMID 41372813
- [Derived] Stromberg S, Baxter BA, Dooley G, LaVergne SM, Gallichotte E, Dutt T, Tipton M, Berry K, Haberman J, Natter N, Webb TL, McFann K, Henao-Tamayo M, Ebel G, Rao S, Dunn J, Ryan EP. Relationships between plasma fatty acids in adults with mild, moderate, or severe COVID-19 and the development of post-acute sequelae. Front Nutr. 2022 Sep 14;9:960409. doi: 10.3389/fnut.2022.960409. eCollection 2022. PMID 36185653
- [Derived] LaVergne SM, Stromberg S, Baxter BA, Webb TL, Dutt TS, Berry K, Tipton M, Haberman J, Massey BR, McFann K, Alnachoukati O, Zier L, Heacock T, Ebel GD, Henao-Tamayo M, Dunn J, Ryan EP. A longitudinal SARS-CoV-2 biorepository for COVID-19 survivors with and without post-acute sequelae. BMC Infect Dis. 2021 Jul 13;21(1):677. doi: 10.1186/s12879-021-06359-2. PMID 34256735